CLINICAL TRIAL: NCT06391918
Title: A Phase 1 Study of GEN2 in Adult Patients With Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: Phase 1 Study of GEN2 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GenVivo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol GVO-1102
Record Dates: First submitted 2024-04-19; First posted 2024-04-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: GEN2 + Valganciclovir — Gene therapy vector product

SUMMARY:
Protocol GVO-1102 is a phase 1, open label, multi-center study in adult patients with locally advanced or metastatic solid tumors. This study includes two parts: dose escalation and dose expansion. In the dose escalation phase, GEN2 will be administered at increasing dose levels via intravenous infusion or intratumoral injection on Days 1, 3 and 8 every 4 weeks. Valganciclovir will start dosing on Day 12 and continue for 10 days (through Day 21). Once a recommended dose has been defined in approximately 35-45 patients, the dose expansion phase will initiate to further assess intravenous administration of GEN2 in specific tumor types. Approximately 15 patients per tumor type will be enrolled in the intravenous dose expansion phase.

DETAILED DESCRIPTION:
GEN2 is a non-replicating off-the-shelf gene therapy vector product being developed as a cancer immunotherapy to activate a patient's immune system against their personal cancer antigens (neoantigens). The vector payload encodes for a suicide gene, an enhanced viral thymidine kinase enzyme (HSV-eTK), which in the presence of a prodrug, valganciclovir, causes the tumor to release patient specific tumor antigens. These neoantigens in the presence of a human immune modulator cytokine, granulocyte-macrophage colony-stimulating factor (hGM-CSF), results in the generation of immune effector cells. These effector cells maintain continually amplifying therapeutic immune responses as more tumor cells are killed and release antigen and will potentially kill any new tumor metastases that arise.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a locally advanced or metastatic solid tumor that has progressed or was non-responsive to prior therapy
* Measurable disease as determined by response evaluation criteria in solid tumors (RECIST) v1.1.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 - 1.
* For patients with HCC: Child-Pugh Class A
* Available archived tumor tissue sample or a lesion that can be safely biopsied if the archived sample is not available.
* Adequate renal, liver and bone marrow function.
* Ability to swallow VGCV tablets.
* Willingness of men and women of child-bearing potential (WCBP) to observe conventional and highly effective birth control for the duration of treatment and for 12 months following the last dose of study treatment. Patients who are pregnant or lactating are excluded.
* For the dose expansion phase: Patients with hepatocellular carcinoma or cutaneous malignancy: no more than 2 prior systemic regimens for metastatic disease. Patients with breast cancer: no more than 2 prior cytotoxic regimens for metastatic disease (single-agent hormone therapy or hormone-based doublets do not count). Patients with cutaneous malignancies includes patients with melanoma, cutaneous squamous cell carcinoma, basal cell carcinoma and Merkel cell carcinoma.
* For the intratumoral injection dose escalation phase: patients with cutaneous malignancy, including patients with melanoma, cutaneous squamous cell carcinoma, basal cell carcinoma and Merkel cell carcinoma. Patients must have at least 1 measurable and injectable lesion and an additional site of measurable distant metastases for assessment of systemic immune response to therapy. Patients may not have received prior treatment with oncolytic therapy. Patients for whom tyrosine kinase inhibitor therapy would be considered standard of care should have received these agents prior to enrollment in this trial. Patients may not have a history of significant bleeding diathesis.

Exclusion Criteria:

* Investigational agent or anticancer therapy within 28 days or 5 elimination half-lives prior to Cycle 1 Day 1.
* Prior receipt of talimogene laherparepvec (TVEC) or any other oncolytic virus (including but not limited to RP1, RP2, or BNT111).; prior receipt of a live vaccine within 28 days prior to Cycle 1 Day 1.
* Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of enrollment (alopecia and other nonacute toxicities are not exclusionary)
* Washout from prior major surgery and radiotherapy (less than 28 days)
* Symptomatic primary central nervous system (CNS) tumor or metastases; symptomatic leptomeningeal carcinomatosis; untreated spinal cord compression. Patients with CNS lesions may be eligible if CNS lesions are asymptomatic or if neurological symptoms are stable, the patient is not receiving steroids to manage CNS symptoms, and no CNS surgery or radiation has been performed for 28 days (14 days for stereotactic radiation).
* Active uncontrolled systemic bacterial, viral, or fungal infection, which in the opinion of the Investigator makes it undesirable for the patient to participate in the trial
* Clinically significant active malabsorption syndrome or other conditions such as refractory nausea and vomiting, external biliary shunt, or significant bowel resection likely to affect gastrointestinal absorption of valganciclovir
* Known contraindications to the ganciclovir class
* For patients with hepatocellular carcinoma, patients with active hepatitis B are excluded; patients with evidence of prior exposure who have a negative hepatitis surface antigen (HbsAg) and who do not require antiviral therapy are allowed. Patients with hepatitis C are allowed but may not be on antiviral therapy during study participation and for two weeks prior to Cycle 1 Day 1.
* Known HIV positivity
* Current treatment with systemic steroids at or above 10 mg/day of prednisone (or its equivalent). Inhalational and topical steroids are acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Determine the recommended phase 2 dose (RP2D) of GEN2 by intravenous infusion and intratumoral injection. | First 28 days.
  The RP2D will be determined by evaluating the number of subjects with treatment related adverse events and Dose Limiting Toxicities

SECONDARY OUTCOMES:
Safety and tolerability as assessed by adverse event monitoring | Up to 24 months
  Adverse events as characterized by type, frequency, severity (graded by NCI CTCAE v 5.0), timing, seriousness and relationship to study therapy
Pharmacokinetics (PK) - Intravenous Administration Cohorts Only: area under the concentration-time curve from the time of dosing to 48 hours after dosing (AUC48h) | Up to 24 months
  AUC48h will be recorded from the PK plasma samples collected
PK - Intravenous Administration Cohorts Only: Maximum Concentration (Cmax) | Up to 24 months
  Cmax will be recorded from the PK plasma samples collected.
To assess replication competent retrovirus (RCR) in peripheral blood mononuclear cells (PBMCs) | Up to 36 months
To assess vector integration into genomic deoxyribonucleic acid (DNA) of PBMCs | Up to 36 months
Overall response rate (ORR) by RECIST 1.1 (Response Evaluation in Solid Tumors Version 1.1) by Investigator Review | Up to 24 months
  ORR is defined as the proportion of participants whose best overall response with confirmation status is rated as (confirmed or unconfirmed) complete response (CR) or (confirmed or unconfirmed) partial response (PR) based on RECIST v1.1.
Disease control rate including a best overall response of Complete Response (CR), Partial Response (PR) or stable disease (SD) | Up to 24 months
  DCR is defined as the proportion of participants whose best overall response with confirmation status is rated as (confirmed or unconfirmed) CR, (confirmed or unconfirmed) PR or stable disease (SD) based on RECIST v1.1.
Duration of response (DOR) | Up to 24 months
  DOR is measured from the day the criteria are first met for time point overall response rated as CR or PR (whichever is first recorded) until the first date of documented radiological disease progression per RECIST v1.1 or death in the absence of progression.
Assess the immunogenicity of GEN2 | Up to 24 months
  Serial blood samples will be screened for anti-vector antibodies (AVAs) and neutralizing antibodies

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - University of Southern California-Keck School of Medicine, Los Angeles, California
  - UCLA Hematology-Oncology, Los Angeles, California
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Iowa Health Care, Iowa City, Iowa
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of Last Patient off.